CLINICAL TRIAL: NCT02328547
Title: Randomized, Double-blinded, Placebo-controlled Trial of Fecal Microbiota Transplantation (FMT) for Diarrhea-Predominant Irritable Bowel Syndrome (IBS-D)
Brief Title: Fecal Microbiota Transplantation for the Treatment of Diarrhea-Predominant Irritable Bowel Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Principal Investigator, Olga Aroniadis, M.D., Montefiore Medical Center
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2014-3941
Record Dates: First submitted 2014-12-16; First posted 2014-12-31 (Estimated); Results first posted 2019-07-02 (Actual); Last update posted 2019-07-02 (Actual); Status verified 2019-06

CONDITIONS: Irritable Bowel Syndrome
Keywords: fecal microbiota transplantation; diarrhea-predominant
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- FMT capsules (Experimental): Intervention: Fecal microbiota transplantation capsules containing extensively screened donor stool, prepared by OpenBiome, Medford, MA. 25 FMT capsules will be take on three consecutive days.
  Interventions: Drug: Fecal microbiota transplantation capsules
- Placebo capsules (Placebo Comparator): Intervention: Placebo capsules that do not contain donor stool or any active drug, prepared by OpenBiome, Medford, MA. 25 placebo capsules will be taken on three consecutive days.
  Interventions: Drug: Placebo capsules

INTERVENTIONS:
Drug: Fecal microbiota transplantation capsules — Fecal microbiota transplantation capsules contain extensively screened donor stool and are prepared by OpenBiome, Medford, MA.
  Other Names: FMT oral capsules
  Arms: FMT capsules
Drug: Placebo capsules — Placebo capsules prepared by OpenBiome, Medford, MA
  Arms: Placebo capsules

SUMMARY:
The objectives of this study are (1) to determine the efficacy of fecal microbiota transplantation (FMT), given as oral capsules, compared with placebo for the treatment of refractory diarrhea-predominant irritable bowel syndrome (IBS-D); (2) determine the impact of FMT on the intestinal microbiome of patients with IBS-D; and (3) assess the safety, feasibility, and tolerability of FMT for patients with IBS-D.

DETAILED DESCRIPTION:
This is a multicenter study including Montefiore Medical Center, Concorde Medical Group PLLC and the Medical Research Center of Connecticut/Yale-New Haven Hospital Langone Medical Center. Patients with IBS-D will be recruited from outpatient gastroenterology clinics at these institutions and referrals from the medical community.

FMT capsules and placebo capsules, provided by OpenBiome, Medford, MA, will be used for this study. Patients will be randomized to undergo FMT using fecal capsules (experimental group) or placebo capsules (control group) via a computer-generated program. All patients will cross-over into the alternate arm of the study at 12 weeks. Therefore, all patients enrolled will receive the experimental drug during the course of the study. Each patient will be enrolled in the study for a total of 6 months.

Intestinal microbiome analyses using DNA sequencing and non-cultivation-based approaches (16S DNA technology) will be performed in all patients in the experimental and control groups to assess stability of the microbiome over time.

ELIGIBILITY:
Inclusion Criteria:

* age 19-65 years
* established diagnosis of IBS-D as determined by Rome III Criteria
* moderate-severe disease activity (as determined by an IBS-Symptom Severity Score ≥175)
* persistent symptoms despite conventional therapy
* normal colonoscopy with biopsies in the past for work-up of IBS symptoms
* negative work-up for celiac disease either by duodenal biopsies or negative serologies

Exclusion Criteria:

* pregnancy
* nursing
* cognitive impairment or severe neuropsychiatric comorbidities who are incapable of providing their own informed consent
* severely immunocompromised or immunosuppressed patients (e.g., organ transplant recipients, severe neutropenia with an absolute neutrophil count of <500cells/mL, current treatment or treatment within 3 months with anti-neoplastic agents and HIV-positive patients with CD4 counts <200cells/mm^3)
* treated with any antibiotics in the 3 months prior to FMT
* GI symptoms can be explained by the presence of an underlying organic disease including, underlying inflammatory bowel disease, infectious enteritis, previously established and untreated small intestinal bacterial overgrowth or known motility disorder
* previous FMT
* severe (anaphylactic) food allergy
* unable to comply with protocol requirements
* American Society of Anesthesiologists (ASA) Physical Status classification IV and V
* acute illness or fever on the day of planned FMT will be excluded (not randomized) with the option of including that subject at a future date
* new antidepressant started or dose of antidepressant change <3 months prior to enrollment
* elevated ESR or CRP within the past 3 months
* baseline laboratory abnormalities on CBC, chemistry or liver tests
* pain score >75 on IBS-SSS

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2018-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Olga C Aroniadis, MD, Principal Investigator — Montefiore Medical Center; Lawrence J Brandt, MD, Principal Investigator — Montefiore Medical Center
Locations (3):
- United States (3):
  - Medical Research Center of Connecticut, Hamden, Connecticut
  - Concorde Medical Group, New York, New York
  - Montefiore Medical Center, The Bronx, New York

REFERENCES:
- [Derived] Aroniadis OC, Brandt LJ, Oneto C, Feuerstadt P, Sherman A, Wolkoff AW, Kassam Z, Sadovsky RG, Elliott RJ, Budree S, Kim M, Keller MJ. Faecal microbiota transplantation for diarrhoea-predominant irritable bowel syndrome: a double-blind, randomised, placebo-controlled trial. Lancet Gastroenterol Hepatol. 2019 Sep;4(9):675-685. doi: 10.1016/S2468-1253(19)30198-0. Epub 2019 Jul 17. PMID 31326345

RESULTS

PARTICIPANT FLOW:
Groups:
- Fecal Microbiota Transplantation Capsules First, Then Placebo: Intervention: 25 Fecal Microbiota Transplantation (FMT) capsules were administered on each of three consecutive days (Day 1, Day 2, Day 3). Patients were seen on Day 10, Week 4, Week 8, and Week 12 after FMT administration. Patients were crossed-over into the Placebo arm at 12 weeks. After cross-over, patients were administered 25 Placebo capsules, that did not contain donor stool or active drug, on each of three consecutive days (Day 1, Day 2, Day 3). Patients were seen on Day 10, Week 4, Week 8, and Week 12 after Placebo dosing. The overall duration of the study was 6 months.
  FMT capsules contained extensively screened donor stool and are prepared by OpenBiome. Placebo capsules contained saline and glycerol. Both FMT and Placebo capsules were prepared by OpenBiome, Medford, MA.
- Placebo Capsules First, Then Fecal Microbiota Transplantation: Intervention: 25 Placebo capsules, that did not contain donor stool or active drug, were administered on each of three consecutive days (Day 1, Day 2, Day 3). Patients were seen on Day 10, Week 4, Week 8, and Week 12 after Placebo administration. Patients were then crossed-over into the FMT arm at 12 weeks. After cross-over, patients were administered 25 Fecal Microbiota Transplantation (FMT) capsules on each of three consecutive days (Day 1, Day 2, Day 3). Patients were seen on Day 10, Week 4, Week 8, and Week 12 after FMT administration. The overall duration of the study was 6 months.
  FMT capsules contained extensively screened donor stool and are prepared by OpenBiome. Placebo capsules contained saline and glycerol. Both FMT and Placebo capsules were prepared by OpenBiome, Medford, MA.
Period: First Intervention (12 Weeks)
Arm/Group | Fecal Microbiota Transplantation Capsules First, Then Placebo | Placebo Capsules First, Then Fecal Microbiota Transplantation
Started | 25 | 23
Completed | 22 | 23
Not Completed | 3 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 2 | 0
Period: Second Intervention (12 Weeks)
Arm/Group | Fecal Microbiota Transplantation Capsules First, Then Placebo | Placebo Capsules First, Then Fecal Microbiota Transplantation
Started | 22 | 23
Completed | 22 | 23
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Fecal Microbiota Transplantation Capsules First, Then Placebo: Intervention: 25 Fecal Microbiota Transplantation (FMT) capsules were administered on each of three consecutive days (Day 1, Day 2, Day 3), then patients were followed for 12 weeks. At 12 weeks, patients crossed over into the alternate arm and received placebo capsules on each of three consecutive days (Day 1, Day 2, Day 3). At 12 weeks, patients crossed over into the alternate arm and received placebo capsules on each of three consecutive days (Day 1, Day 2, Day 3).
  FMT capsules contained extensively screened donor stool and are prepared by OpenBiome. Placebo capsules contained saline and glycerol. Both FMT and Placebo capsules were prepared by OpenBiome, Medford, MA.
- Placebo Capsules First, Then Fecal Microbiota Transplantation: Intervention: 25 Placebo capsules, that did not contain donor stool or active drug, were administered on each of three consecutive days (Day 1, Day 2, Day 3), then patients were followed for 12 weeks. At 12 weeks, patients crossed over into the alternate arm and received fecal microbiota transplantation capsules on each of three consecutive days (Day 1, Day 2, Day 3).
  FMT capsules contained extensively screened donor stool and are prepared by OpenBiome. Placebo capsules contained saline and glycerol. Both FMT and Placebo capsules were prepared by OpenBiome, Medford, MA.
- Total: Total of all reporting groups
Arm/Group | Fecal Microbiota Transplantation Capsules First, Then Placebo | Placebo Capsules First, Then Fecal Microbiota Transplantation | Total
Number analyzed (Participants) | 25 | 23 | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.8 (12.3) | 39.0 (11.7) | 38.4 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 9 | 18
  Male | 16 | 14 | 30
Race (NIH/OMB) [Count of Participants; unit: Participants] — 'More than one race' category identified as "Other" in study data
  Participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 2 | 2 | 4
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 0 | 0 | 0
    White | 21 | 19 | 40
    More than one race | 2 | 2 | 4
    Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 25 | 23 | 48
IBS-SSS [Mean (Standard Deviation); unit: units on a scale] — Irritable Bowel Syndrome-Symptom Severity Score (IBS-SSS) is measured on a scale range of 0-500 (min-max) via administration of a questionnaire. Higher scores are indicative of greater disease severity of symptoms based on a validated method. Subjects are categorized as having mild (75-175), moderate (175-300), or severe (>300) irritable bowel syndrome (IBS) based on symptomology.
  units on a scale | 282 (65) | 309 (64) | 294 (65)
IBS-QOL [Mean (Standard Deviation); unit: units on a scale] — Irritable Bowel Syndrome-Quality of Life (IBS-QOL) is administered via a questionnaire of 34 items each with an individual five-point response scale. The responses to these items are summed and averaged for a total score and then transformed to a 100-point scale for ease of interpretation based on a validated method. IBS-QOL is measured on a scale range of 0-100. Higher IBS-QOL scores are indicative of a better IBS-specific quality of life.
  units on a scale | 53 (18) | 52 (18) | 52 (18)
Hospital Anxiety and Depression Scale (HADS). HADS-A (Anxiety) [Mean (Standard Deviation); unit: units on a scale] — The Hospital Anxiety and Depression Scale (HADS) is a fourteen item scale which is administered via questionnaire. Seven of the items relate to anxiety and seven relate to depression. Each item on the questionnaire is scored from 0-3 and this means that a person can score between 0 and 21 for either anxiety or depression. The HADS uses a scale and therefore the data returned from the HADS is ordinal. Higher HADS scores are indicative of more severe depression and anxiety.
  HADS-A (Anxiety component)
  units on a scale | 8.3 (4.7) | 7.2 (3.6) | 7.8 (4.2)
Hospital Anxiety and Depression Scale (HADS) HADS-D (Depression) [Mean (Standard Deviation); unit: units on a scale] — The Hospital Anxiety and Depression Scale (HADS) is a fourteen item scale which is administered via questionnaire. Seven of the items relate to anxiety and seven relate to depression. Each item on the questionnaire is scored from 0-3 and this means that a person can score between 0 and 21 for either anxiety or depression. The HADS uses a scale and therefore the data returned from the HADS is ordinal. Higher HADS scores are indicative of more severe depression and anxiety.
  HADS-D (Depression component)
  units on a scale | 4.6 (4.3) | 5.1 (3.0) | 4.8 (3.7)
Bristol Stool Form Scale (BSFS) [Mean (Standard Deviation); unit: units on a scale] — The Bristol Stool Form Scale is administered via questionnaire. This scale is a diagnostic medical tool designed to classify the form of human feces into seven categories. Assigned categories range from 1-7 based on appearance of the stool. Type 1 and 2 stools indicate constipation. Type 4 are the ideal stools as they are easy to defecate while not containing excess liquid, Type 5 tends towards diarrhea, and Types 6 and 7 indicate diarrhea.
  units on a scale | 5.0 (0.8) | 6.0 (0.9) | 6.0 (0.9)

OUTCOME MEASURES:

1. Primary Outcome: Within and Between Group Comparisons of Disease Severity as Determined by Irritable Bowel Syndrome-Symptom Severity Score (IBS-SSS)
Description: Within and between group comparisons of changes (from baseline) in Irritable Bowel Syndrome-Symptom Severity Score (IBS-SSS), obtained via administration of a Questionnaire, for each of the two arms/groups (FMT capsules first, and placebo capsules first). The scale range was 0-500 (min-max). Scores were averaged among time points to yield an overall mean score. Higher scores were indicative of greater disease severity (worse outcome). Subjects were categorized as having mild (75-175), moderate (175-300), or severe (>300) irritable bowel syndrome (IBS) based on symptomology.
  Only the following time points were analyzed: Baseline vs Week 12 and Week 24.
Time Frame: Baseline, Week 12 (before cross-over), Week 24
Population: Participants were randomized to FMT first followed by placebo (n=25) OR to placebo first followed by FMT (n=23) and analyzed in these groups. Participants who received FMT 1st and those who received FMT 2nd were not pooled together into one group because of potential carry-over effects.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- FMT Capsules, Followed by Placebo Capsules: Intervention: 25 fecal microbiota transplantation (FMT) capsules were administered on each of three consecutive days (Day 1, Day 2, Day 3), then patients were followed for 12 weeks. At 12 weeks, patients crossed over into the alternate arm and received placebo capsules on each of three consecutive days (Day 1, Day 2, Day 3). Analyses included change in outcome measure between baseline and 12 weeks.
- Placebo Capsules, Followed by FMT Capsules: Intervention: 25 placebo capsules were administered on each of three consecutive days (Day 1, Day 2, Day 3), then patients were followed for 12 weeks. At 12 weeks, patients crossed over into the alternate arm and received fecal microbiota transplantation capsules on each of three consecutive days (Day 1, Day 2, Day 3). Analyses included change in outcome measure between baseline and 12 weeks.
Arm/Group | FMT Capsules, Followed by Placebo Capsules | Placebo Capsules, Followed by FMT Capsules
Number analyzed (Participants) | 25 | 23
units on a scale
  Baseline | 282 (65) | 309 (64)
  Week 12 | 221 (105) | 236 (95)
  Week 24 | 208 (111) | 157 (101)

2. Secondary Outcome: Within and Between Group Comparisons of Quality of Life as Determined by the Irritable Bowel Syndrome-Quality of Life (IBS-QOL) Score
Description: Within and between group comparisons of changes (from baseline) in Irritable Bowel Syndrome-Quality of Life (IBS-QOL), obtained via administration of a Questionnaire, for each of the two arms/groups (FMT capsules first, and placebo capsules first). Irritable Bowel Syndrome-Quality of Life (IBS-QOL) is administered via a questionnaire of 34 items each with an individual five-point response scale. The responses to these items are summed and averaged for a total score and then transformed to a 100-point scale for ease of interpretation based on a validated method. IBS-QOL is measured on a scale range of 0-100. Higher IBS-QOL scores are indicative of a better IBS-specific quality of life.
  Only the following time points were analyzed: Baseline vs Week 12
Time Frame: Baseline, Week 12 (before cross-over), Week 24
Population: Participants were randomized to FMT first followed by placebo (n=25) OR to placebo first followed by FMT (n=23) and analyzed in these groups. Participants who received FMT 1st and those who received FMT 2nd were not pooled together into one group because of potential carry-over effects. As such, data for crossover intervention couldn't be reported.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | FMT Capsules, Followed by Placebo Capsules | Placebo Capsules, Followed by FMT Capsules
Number analyzed (Participants) | 25 | 23
units on a scale
  Baseline | 53 (18) | 52 (18)
  Week 12 | 65 (18) | 66 (17)
  Week 24 | 70 (18) | 76 (17)

3. Secondary Outcome: Intestinal Microbiota Composition Pre- and Post-FMT (Fecal Microbiota Transplantation)
Description: Microbiota composition before and after FMT were assessed among FMT responders and FMT non-responders. Only patients who received FMT capsules at the start of this clinical trial were included. Placebo capsule recipients were not included in these analyses. Data were analyzed up to 12 weeks and not beyond. Microbiome data following cross-over were not analyzed because of the potential for carry-over and order effects in the second half of the trial.
  Outcomes assessed included alpha and beta diversity (Jensen-Shannon divergence) and abundance of Bacteroidetes, Firmicutes and Prevotella. All of the microbiome data that were analyzed are included in the table below. No additional microbiome data from this clinical trial were analyzed.
Time Frame: Baseline, Week 1, Week 4 and Week 12
Measure: Mean (Standard Deviation); unit: percentage of bacteria
Groups:
- FMT Responders: Includes patients who received FMT capsules at the start of the clinical trial and who responded to FMT. FMT response was defined as a decrease of at least 50 points in the IBS-SSS at week 12 compared with baseline score.
- FMT Non-responders: Includes patients who received FMT capsules at the start of the clinical trial but who did not respond to FMT. FMT non-response was defined as a less than 50 point decrease in the IBS-SSS at week 12 compared with baseline score.
Arm/Group | FMT Responders | FMT Non-responders
Number analyzed (Participants) | 11 | 11
percentage of bacteria
  Bacteroidetes - Baseline | 0.41 (0.19) | 0.35 (0.10)
  Bacteroidetes - Week 1 | 0.43 (0.15) | 0.34 (0.10)
  Bacteroidetes - Week 4 | 0.38 (0.14) | 0.34 (0.09)
  Bacteroidetes - Week 12 | 0.47 (0.14) | 0.34 (0.10)

4. Secondary Outcome: Anxiety as Measured by the Hospital Anxiety and Depression Scale (HADS). HADS-A (Anxiety)
Description: Anxiety at baseline and at the time of cross-over (Week 12) as measured by Hospital Anxiety and Depression Scale (HADS). HADS-A (Anxiety)
  The Hospital Anxiety and Depression Scale (HADS) is a fourteen item scale which was administered via questionnaire. Seven of the items relate to anxiety (HADS-A) and seven relate to depression (HADS-D). Each item on the questionnaire is scored from 0-3 and this means that a person can score between 0 and 21 for either anxiety or depression. The HADS uses a scale and therefore the data returned from the HADS is ordinal. Higher HADS scores are indicative of more severe depression and anxiety.
  Only the following time points were analyzed: Baseline vs Week 12
Time Frame: Baseline, Week 12 (before cross-over), Week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | FMT Capsules, Followed by Placebo Capsules | Placebo Capsules, Followed by FMT Capsules
Number analyzed (Participants) | 25 | 23
score on a scale
  Baseline | 8.3 (4.7) | 7.2 (3.6)
  Week 12 | 8.6 (5.0) | 7.4 (4.6)
  Week 24 | 7.9 (4.8) | 5.6 (3.6)

5. Secondary Outcome: Depression as Measured by the Hospital Anxiety and Depression Scale (HADS). HADS-D (Depression)
Description: Depression at baseline and at the time of cross-over (Week 12) as measured by Hospital Anxiety and Depression Scale (HADS). HADS-D (Depression)
  The Hospital Anxiety and Depression Scale (HADS) is a fourteen item scale which was administered via questionnaire. Seven of the items relate to anxiety (HADS-A) and seven relate to depression (HADS-D). Each item on the questionnaire is scored from 0-3 and this means that a person can score between 0 and 21 for either anxiety or depression. The HADS uses a scale and therefore the data returned from the HADS is ordinal. Higher HADS scores are indicative of more severe depression and anxiety.
  Only the following time points were analyzed: Baseline vs Week 12
Time Frame: Baseline, Week 12 (before cross-over), Week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | FMT Capsules, Followed by Placebo Capsules | Placebo Capsules, Followed by FMT Capsules
Number analyzed (Participants) | 25 | 23
score on a scale
  Baseline | 4.6 (4.3) | 5.1 (3.0)
  Week 12 | 4.0 (4.1) | 4.0 (2.6)
  Week 24 | 3.8 (3.5) | 3.4 (2.8)

6. Secondary Outcome: Bowel Consistency as Measured by the Bristol Stool Form Scale (BSFS)
Description: Bowel consistency as measured by the Bristol Stool Form Scale on a daily basis.
  The Bristol Stool Form Scale was administered via questionnaire. This scale is a diagnostic medical tool designed to classify the form of human feces into seven categories. Assigned categories range from 1-7 based on appearance of the stool. Type 1 and 2 stools indicate constipation. Type 4 are the ideal stools as they are easy to defecate while not containing excess liquid, Type 5 tends towards diarrhea, and Types 6 and 7 indicate diarrhea.
  Only the following time points were analyzed: Baseline vs Week 12
Time Frame: Baseline, Week 12 (before cross-over), Week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | FMT Capsules, Followed by Placebo Capsules | Placebo Capsules, Followed by FMT Capsules
Number analyzed (Participants) | 25 | 23
score on a scale
  Baseline | 5 (0.8) | 6 (0.9)
  Week 12 | 4 (1.0) | 5 (1.1)
  Week 24 | 4 (1.0) | 4 (1.3)

7. Secondary Outcome: Number of Participants With Adverse Events as a Measure of Safety and Tolerability
Description: The total number of participants in each of the arms/groups (FMT and Placebo) who experienced at least one adverse event (AE) as recorded in patient diaries.
Time Frame: All AEs over 24 weeks
Population: Participants were randomized to FMT first followed by placebo (n=25) OR to placebo first followed by FMT (n=23) and analyzed in these groups. Participants who received FMT 1st and those who received FMT 2nd were pooled together into one group.
Measure: Count of Participants; unit: Participants
Groups:
- FMT Capsules: Intervention: 25 fecal microbiota transplantation (FMT) capsules were administered on each of three consecutive days (Day 1, Day 2, Day 3) either at the start of the trial or at cross-over (week 12).
- Placebo Capsules: Intervention: 25 placebo capsules were administered on each of three consecutive days (Day 1, Day 2, Day 3) at the start of the trial or at cross-over (week 12).
Arm/Group | FMT Capsules | Placebo Capsules
Number analyzed (Participants) | 48 | 48
Participants
  Any Adverse Event | 23 | 24
  No Adverse Events | 25 | 24

8. Secondary Outcome: Satisfaction With Fecal Microbiota Transplantation (FMT)
Description: Weekly assessments of satisfaction with the Fecal Microbiota Transplantation (FMT) will be recorded in patient diaries.
Time Frame: Week 12 following administration of FMT
Population: Data was not collected and, therefore, the outcome cannot be reported.
Groups:
- FMT Capsules, Followed by Placebo Capsules: Intervention: 25 fecal microbiota transplantation (FMT) capsules were administered on each of three consecutive days (Day 1, Day 2, Day 3), then patients were followed for 12 weeks. At 12 weeks, patients crossed over into the alternate arm and received placebo capsules on each of three consecutive days (Day 1, Day 2, Day 3).
- Placebo Capsules, Followed by FMT Capsules: Intervention: 25 placebo capsules were administered on each of three consecutive days (Day 1, Day 2, Day 3), then patients were followed for 12 weeks. At 12 weeks, patients crossed over into the alternate arm and received fecal microbiota transplantation capsules on each of three consecutive days (Day 1, Day 2, Day 3).
Arm/Group | FMT Capsules, Followed by Placebo Capsules | Placebo Capsules, Followed by FMT Capsules
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Change in Bowel Habits and Abdominal Pain After Fecal Microbiota Transplantation (FMT)
Description: Degree of improvement in bowel habits and abdominal pain will be recorded in patient diaries.
Time Frame: Week 12 following administration of FMT
Population: Data was not collected and, therefore, the outcome cannot be reported.
Arm/Group | FMT Capsules, Followed by Placebo Capsules | Placebo Capsules, Followed by FMT Capsules
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Number of Doctor or Emergency Department (ED) Visits Post-Fecal Microbiota Transplantation (Post-FMT) for Irritable Bowel Syndrome-D (IBS-D) Related Symptoms
Description: The number of doctor or ED visits post-Fecal Microbiota Transplantation for Irritable Bowel Syndrome-D (IBS-D) related symptoms will be recorded in patient diaries.
Time Frame: Week 12 following administration of FMT
Population: Data was not collected and, therefore, the outcome cannot be reported.
Arm/Group | FMT Capsules, Followed by Placebo Capsules | Placebo Capsules, Followed by FMT Capsules
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Initiation of New Medications Post-FMT for the Treatment of IBS-D Symptoms
Description: Initiation of new medications post-FMT for the treatment of IBS-D symptoms will be recorded in patient diaries.
Time Frame: Week 12 following administration of FMT
Population: Data was not collected and, therefore, the outcome cannot be reported.
Arm/Group | FMT Capsules, Followed by Placebo Capsules | Placebo Capsules, Followed by FMT Capsules
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Patient Attitudes Towards Fecal Microbiota Transplantation (FMT)
Description: Patient attitudes towards Fecal Microbiota Transplantation (FMT) will be recorded in patient diaries.
Time Frame: Week 12 following administration of FMT
Population: Data was not collected and, therefore, the outcome cannot be reported.
Arm/Group | FMT Capsules, Followed by Placebo Capsules | Placebo Capsules, Followed by FMT Capsules
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Tolerability of Fecal Microbiota Transplantation (FMT)
Description: Tolerability of Fecal Microbiota Transplantation (FMT) will be maintained in patient diaries.
Time Frame: Week 12 following administration of FMT
Population: Data was not collected and, therefore, the outcome cannot be reported.
Arm/Group | FMT Capsules, Followed by Placebo Capsules | Placebo Capsules, Followed by FMT Capsules
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: Intestinal Microbiota Composition Pre- and Post-FMT (Fecal Microbiota Transplantation)
Description: Microbiota composition before and after FMT were assessed among FMT responders and FMT non-responders. Only patients who received FMT capsules at the start of this clinical trial were included. Placebo capsule recipients were not included in these analyses. Data were analyzed up to 12 weeks and not beyond. Microbiome data following cross-over were not analyzed because of the potential for carry-over and order effects in the second half of the trial.
  Outcomes assessed included alpha and beta diversity (Jensen-Shannon divergence) and abundance of Bacteroidetes, Firmicutes and Prevotella. All of the microbiome data that were analyzed are included in the table below. No additional microbiome data from this clinical trial were analyzed.
  The Alpha Diversity Index is a quantitative measure that reflects the diversity of bacterial species in a sample. The greater the index, the more diverse the intestinal microbiota.
Time Frame: Baseline, Week 1, Week 4 and Week 12
Measure: Mean (Standard Deviation); unit: index
Arm/Group | FMT Responders | FMT Non-responders
Number analyzed (Participants) | 11 | 11
index
  Alpha Diversity - Baseline | 3.96 (0.43) | 4.16 (0.41)
  Alpha-Diversity - Week 1 | 4.00 (0.41) | 4.13 (0.28)
  Alpha Diversity - Week 4 | 4.05 (0.59) | 4.29 (0.29)
  Alpha Diversity - Week 12 | 4.02 (0.62) | 4.29 (0.29)

15. Secondary Outcome: Intestinal Microbiota Composition Pre- and Post-FMT (Fecal Microbiota Transplantation)
Description: Microbiota composition before and after FMT were assessed among FMT responders and FMT non-responders. Only patients who received FMT capsules at the start of this clinical trial were included. Placebo capsule recipients were not included in these analyses. Data were analyzed up to 12 weeks and not beyond. Microbiome data following cross-over were not analyzed because of the potential for carry-over and order effects in the second half of the trial.
  Outcomes assessed included alpha and beta diversity (Jensen-Shannon divergence) and abundance of Bacteroidetes, Firmicutes and Prevotella. All of the microbiome data that were analyzed are included in the table below. No additional microbiome data from this clinical trial were analyzed.
  The Beta Diversity Index or Jensen-Shannon divergence is a quantitative measure that reflects the diversity of bacterial species between two different regions. The greater the index, the more diverse the intestinal microbiota between the two regions.
Time Frame: Baseline, Week 1, Week 4 and Week 12
Measure: Mean (Standard Deviation); unit: index
Arm/Group | FMT Responders | FMT Non-responders
Number analyzed (Participants) | 11 | 11
index
  Jensen-Shannon Diversity - Baseline | 0.52 (0.12) | 0.48 (0.22)
  Jensen-Shannon Diversity - Week 1 | 0.44 (0.16) | 0.40 (0.16)
  Jensen Shannon Diversity - Week 4 | 0.43 (0.14) | 0.38 (0.16)
  Jensen Shannon Diversity - Week 12 | 0.41 (0.16) | 0.40 (0.15)

16. Secondary Outcome: Intestinal Microbiota Composition Pre- and Post-FMT (Fecal Microbiota Transplantation)
Description: as for outcome 3
Time Frame: Baseline, Week 1, Week 4 and Week 12
Measure: Mean (Standard Deviation); unit: percentage of bacteria
Arm/Group | FMT Responders | FMT Non-responders
Number analyzed (Participants) | 11 | 11
percentage of bacteria
  Firmicutes - Baseline | 0.51 (0.19) | 0.55 (0.12)
  Firmicutes - Week 1 | 0.50 (0.15) | 0.54 (0.11)
  Firmicutes - Week 4 | 0.50 (0.13) | 0.57 (0.12)
  Firmicutes - Week 12 | 0.46 (0.12) | 0.56 (0.09)

17. Secondary Outcome: Intestinal Microbiota Composition Pre- and Post-FMT (Fecal Microbiota Transplantation)
Description: Microbiota composition before and after FMT were assessed among FMT responders and FMT non-responders. Only patients who received FMT capsules at the start of this clinical trial were included. Placebo capsule recipients were not included in these analyses. Data were analyzed up to 12 weeks and not beyond. Microbiome data following cross-over were not analyzed because of the potential for carry-over and order effects in the second half of the trial.
  Outcomes assessed included alpha and beta diversity (Jensen-Shannon divergence) and abundance of Bacteroidetes, Firmicutes and Prevotella. All of the microbiome data that were analyzed are included in the table below. No additional microbiome data from this clinical trial were analyzed. Information on abundance of Prevotella was only available at baseline and week 1.
Time Frame: Baseline and Week 1
Measure: Mean (Standard Deviation); unit: percentage of bacteria
Arm/Group | FMT Responders | FMT Non-responders
Number analyzed (Participants) | 11 | 11
percentage of bacteria
  Prevotella - Baseline | 0.12 (0.18) | 0.04 (0.12)
  Prevotella - Week 1 | 0.14 (0.19) | 0.03 (0.09)

ADVERSE EVENTS:
Time Frame: 6 months
Description: Adverse Events (AEs) were solicited during each patient visit. Additionally, patients, were asked to maintain a daily diary of AEs in a specifically dedicated diary developed by the research team to facilitate standardized reporting.
Groups:
- FMT Capsules: 25 Fecal Microbiota Transplantation (FMT) capsules were administered on each of three consecutive days (Day 1, Day 2, Day 3) at initiation of the trial or at the time of cross-over (week 12).
  FMT capsules contained extensively screened donor stool and were prepared by OpenBiome, Medford, MA.
- Placebo Capsules: 25 placebo capsules, that did not contain donor stool or any active drug, were administered on each of three consecutive days (Day 1, Day 2, Day 3) at initiation of the trial or at the time of cross-over (week 12).
  Placebo capsules contained saline and glycerol. ann were prepared by OpenBiome, Medford, MA.
Arm/Group | FMT Capsules | Placebo Capsules
All-Cause Mortality (participants affected / at risk) | 0/48 | 0/48
Serious Adverse Events (participants affected / at risk) | 0/48 | 1/48
Other Adverse Events (participants affected / at risk) | 23/48 | 24/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FMT Capsules (N=48) | Placebo Capsules (N=48)
cholecystectomy (Gastrointestinal disorders) | 0 (0) | 1 (1) — One study-unrelated SAE was reported. This participant underwent cholecystectomy for acute cholecystitis 2 months after ingesting placebo capsules.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | FMT Capsules (N=48) | Placebo Capsules (N=48)
Abdominal Pain (Gastrointestinal disorders) | 5 | 4
Nausea (Gastrointestinal disorders) | 4 | 2
Worsening of Diarrhea (Gastrointestinal disorders) | 3 | 8
Constipation (Gastrointestinal disorders) | 2 | 0
Bloating (Gastrointestinal disorders) | 2 | 5
Regurgitation/Emesis (Gastrointestinal disorders) | 2 | 0
Fatigue (Gastrointestinal disorders) | 2 | 1
Gas (Gastrointestinal disorders) | 1 | 4
Belching (Gastrointestinal disorders) | 1 | 0
Loss of Appetite (Gastrointestinal disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-04-24): https://cdn.clinicaltrials.gov/large-docs/47/NCT02328547/Prot_SAP_000.pdf